CLINICAL TRIAL: NCT00251979
Title: A Randomised, Double-blind, Parallel-group, Placebo Controlled Study of Esomeprazole i.v. (Bolus Infusion of 80 mg Followed by a Continuous Infusion of 8 mg Per Hour) Administered for 72 Hours to Assess Prevention of Rebleeding in Subjects That Have Undergone Successful Primary Endoscopic Haemostasis of a Bleeding Peptic Ulcer - the PUB Study.
Brief Title: A Study to Prevent Rebleeding After Initial Successful Primary Endoscopic Haemostasis of a Bleeding Peptic Ulcer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D961DC00001
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Results first posted 2011-06-17 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-05

CONDITIONS: Gastrointestinal Hemorrhage
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole

SUMMARY:
This study is being carried out to see if constant 3 days infusion of Nexium is effective in preventing rebleeding after an endoscopic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signs of a bleeding in the stomach
* One endoscopically confirmed bleeding ulcer in the stomach or duodenum

Exclusion Criteria:

* Malignancy or other advanced disease.
* Major cardiovascular event.
* Severe hepatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1312 (Actual)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Nexium Medical Sciences Director, Study Director — AstraZeneca; Joseph Sung, MD, Principal Investigator — Chinese University of Hong Kong
Locations (78):
- Austria (6):
  - Research Site, Braunau/Inn
  - Research Site, Feldbach
  - Research Site, Graz
  - Research Site, Krems
  - Research Site, Vienna
  - Research Site, Wels
- Denmark (8):
  - Research Site, Aalborg
  - Research Site, Amager
  - Research Site, Copenhagen
  - Research Site, Glostrup Municipality
  - Research Site, Holstebro
  - Research Site, Odense
  - Research Site, Randers
  - Research Site, Slagelse
- Finland (2):
  - Research Site, Helsinki
  - Research Site, Kuopio
- France (7):
  - Research Site, Amiens
  - Research Site, Bordeaux
  - Research Site, Clermont-Ferrand
  - Research Site, Lille
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Rouen
- Germany (9):
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Celle
  - Research Site, Dresden
  - Research Site, Karlsruhe
  - Research Site, Leipzig
  - Research Site, Ludwigshafen
  - Research Site, Magdeburg
  - Research Site, Weimar
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- Research Site, Hong Kong, Hong Kong
- Netherlands (6):
  - Research Site, Arnhem
  - Research Site, Dordrecht
  - Research Site, Hengelo
  - Research Site, Nieuwegein
  - Research Site, Rotterdam
  - Research Site, Zwolle
- Norway (6):
  - Research Site, Ålesund
  - Research Site, Drammen
  - Research Site, Kristiansand
  - Research Site, Lorenskog
  - Research Site, Oslo
  - Research Site, Tønsberg
- Romania (5):
  - Research Site, Bucharest
  - Research Site, Craiova
  - Research Site, Iași
  - Research Site, Tg. Mures
  - Research Site, Timișoara
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- South Africa (3):
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Pietermaritzburg
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Sabadell
  - Research Site, Santiago
- Sweden (10):
  - Research Site, Gothenburg
  - Research Site, Karlstad
  - Research Site, Kristianstad
  - Research Site, Linköping
  - Research Site, Norrköping
  - Research Site, Östersund
  - Research Site, Skövde
  - Research Site, Stockholm
  - Research Site, Sundsvall
  - Research Site, Trollhättan
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Bursa
  - Research Site, Izmir
  - Research Site, İzmit
- United Kingdom (3):
  - Research Site, Birmingham
  - Research Site, Derby
  - Research Site, Leeds

REFERENCES:
- [Derived] Lau J, Lind T, Persson T, Eklund S. Effect of baseline characteristics on response to proton pump inhibitors in patients with peptic ulcer bleeding. J Dig Dis. 2017 Feb;18(2):99-106. doi: 10.1111/1751-2980.12447. PMID 28070941
- [Derived] Kuipers EJ, Sung JJ, Barkun A, Mossner J, Jensen D, Stuart R, Lau JY, Ahlbom H, Lind T, Kilhamn J. Safety and tolerability of high-dose intravenous esomeprazole for prevention of peptic ulcer rebleeding. Adv Ther. 2011 Feb;28(2):150-9. doi: 10.1007/s12325-010-0095-5. Epub 2010 Dec 15. PMID 21181319
- [Derived] Barkun AN, Adam V, Sung JJ, Kuipers EJ, Mossner J, Jensen D, Stuart R, Lau JY, Naucler E, Kilhamn J, Granstedt H, Liljas B, Lind T. Cost effectiveness of high-dose intravenous esomeprazole for peptic ulcer bleeding. Pharmacoeconomics. 2010;28(3):217-30. doi: 10.2165/11531480-000000000-00000. PMID 20151726
- [Derived] Sung JJ, Barkun A, Kuipers EJ, Mossner J, Jensen DM, Stuart R, Lau JY, Ahlbom H, Kilhamn J, Lind T; Peptic Ulcer Bleed Study Group. Intravenous esomeprazole for prevention of recurrent peptic ulcer bleeding: a randomized trial. Ann Intern Med. 2009 Apr 7;150(7):455-64. doi: 10.7326/0003-4819-150-7-200904070-00105. Epub 2009 Feb 16. PMID 19221370

RESULTS

PARTICIPANT FLOW:
Groups:
- Esomeprazole: Esomeprazole iv for 72 h followed by esomeprazole oral 40 mg od for 27 days
- Placebo: Placebo iv for 72 h followed by esomeprazole oral 40 mg od for 27 days
Period: Overall Study
Arm/Group | Esomeprazole | Placebo
Started | 375 (ITT population) | 389 (ITT population)
Completed | 337 | 349
Not Completed | 38 | 40
Not completed — Protocol Violation | 3 | 5
Not completed — Adverse Event | 11 | 17
Not completed — Withdrawal by Subject | 13 | 7
Not completed — Lost to Follow-up | 8 | 6
Not completed — Death | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole | Placebo | Total
Number analyzed (Participants) | 375 | 389 | 764
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 182 | 210 | 392
  >=65 years | 193 | 179 | 372
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 121 | 242
  Male | 254 | 268 | 522

OUTCOME MEASURES:

1. Primary Outcome: Clinically Significant Rebleeding Within 72 Hours of Continous Infusion of Esomeprazole or Placebo
Time Frame: Within 72 hours
Measure: Number; unit: Participants
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 375 | 389
Participants | 22 | 40

2. Secondary Outcome: Clinically Significant Rebleeding Within 7 Days
Time Frame: Within 7 days
Measure: Number; unit: Participants
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 375 | 389
Participants | 27 | 50

3. Secondary Outcome: Clinically Significant Rebleeding Within 30 Days
Time Frame: Within 30 days
Measure: Number; unit: Participants
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 375 | 389
Participants | 29 | 53

4. Secondary Outcome: Death Within 72 Hours
Time Frame: Within 72 hours
Measure: Number; unit: Participants
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 375 | 389
Participants | 1 | 0

5. Secondary Outcome: Death Within 30 Days
Time Frame: Within 30 days
Measure: Number; unit: Participants
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 375 | 389
Participants | 3 | 8

6. Secondary Outcome: Death Related to Rebleeding Within 30 Days as Judged by the EpC
Time Frame: Within 30 days
Measure: Number; unit: Participants
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 375 | 389
Participants | 2 | 3

7. Secondary Outcome: Requirement for Surgery Within 72 Hours
Time Frame: Within 72 hours
Measure: Number; unit: Participants
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 375 | 389
Participants | 5 | 9

8. Secondary Outcome: Requirement for Surgery Within 30 Days
Time Frame: Within 30 days
Measure: Number; unit: Participants
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 375 | 389
Participants | 10 | 21

9. Secondary Outcome: Requirement for Endoscopic Re-treatment Within 72 Hours
Time Frame: Within 72 hours
Measure: Number; unit: Participants
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 375 | 389
Participants | 16 | 32

10. Secondary Outcome: Requirement for Endoscopic Re-treatment Within 30 Days
Time Frame: Within 30 days
Measure: Number; unit: Participants
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 375 | 389
Participants | 24 | 45

11. Secondary Outcome: Number of Blood Units Transfused Within 72 Hours
Time Frame: Within 72 hours
Measure: Number; unit: blood units
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 375 | 389
blood units | 492 | 738

12. Secondary Outcome: Number of Blood Units Transfused Within 30 Days
Time Frame: within 30 days
Measure: Number; unit: blood units
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 375 | 389
blood units | 589 | 935

13. Secondary Outcome: Number of Days Hospitalized Due to Rebleeding During the 30-day Treatment Period
Time Frame: Within 30 days
Measure: Number; unit: days
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 375 | 389
days | 284 | 500

ADVERSE EVENTS:
Arm/Group | Esomeprazole | Placebo
Serious Adverse Events (participants affected / at risk) | 61 | 68
Other Adverse Events (participants affected / at risk) | 87/375 | 129/389
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Esomeprazole | Placebo
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1/375 | 2/389
ACUTE PSYCHOSIS (Psychiatric disorders) | 1/375 | 0/389
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/375 | 1/389
ANGINA PECTORIS (Cardiac disorders) | 1/375 | 0/389
ANGINA UNSTABLE (Cardiac disorders) | 1/375 | 0/389
ATRIAL FIBRILLATION (Cardiac disorders) | 0/375 | 3/389
BENIGN GASTRIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/375 | 1/389
BRADYCARDIA (Cardiac disorders) | 1/375 | 0/389
CARDIAC FAILURE (Cardiac disorders) | 1/375 | 0/389
CHOLECYSTITIS (Hepatobiliary disorders) | 1/375 | 0/389
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1/375 | 0/389
COLONIC POLYP (Gastrointestinal disorders) | 0/375 | 1/389
CONSTIPATION (Gastrointestinal disorders) | 0/375 | 1/389
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1/375 | 0/389
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1/375 | 0/389
DISCOMFORT (Metabolism and nutrition disorders) | 1/375 | 0/389
DISLOCATION OF JOINT PROSTHESIS (Injury, poisoning and procedural complications) | 1/375 | 0/389
DIZZINESS (Nervous system disorders) | 0/375 | 1/389
DUODENAL PERFORATION (Gastrointestinal disorders) | 0/375 | 1/389
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 16/375 | 21/389
DUODENAL ULCER PERFORATION (Gastrointestinal disorders) | 0/375 | 1/389
ERYSIPELAS (Infections and infestations) | 0/375 | 1/389
FATIGUE (Infections and infestations) | 1/375 | 0/389
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/375 | 1/389
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 7/375 | 13/389
GASTRIC ULCER PERFORATION (Gastrointestinal disorders) | 0/375 | 1/389
GASTROENTERITIS (Infections and infestations) | 1/375 | 0/389
GASTROINTESTINAL ANGIODYSPLASIA HAEMORRHAGIC (Congenital, familial and genetic disorders) | 0/375 | 1/389
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1/375 | 1/389
GASTROINTESTINAL STROMAL TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/375 | 0/389
GOUT (Metabolism and nutrition disorders) | 2/375 | 1/389
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0/375 | 3/389
HAEMOGLOBIN DECREASED (Musculoskeletal and connective tissue disorders) | 0/375 | 1/389
HIP FRACTURE (Injury, poisoning and procedural complications) | 1/375 | 0/389
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0/375 | 1/389
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1/375 | 0/389
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0/375 | 1/389
LUNG INFECTION (Infections and infestations) | 1/375 | 0/389
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0/375 | 1/389
MELAENA (Gastrointestinal disorders) | 2/375 | 0/389
MYOCARDIAL INFARCTION (Cardiac disorders) | 4/375 | 5/389
OSTEOLYSIS (Musculoskeletal and connective tissue disorders) | 1/375 | 0/389
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0/375 | 1/389
PEPTIC ULCER PERFORATION (Gastrointestinal disorders) | 0/375 | 1/389
PERIPHERAL NERVE LESION (Nervous system disorders) | 1/375 | 0/389
PERITONITIS (Gastrointestinal disorders) | 0/375 | 1/389
PHLEBITIS (Vascular disorders) | 1/375 | 0/389
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1/375 | 0/389
PNEUMONIA (Infections and infestations) | 1/375 | 0/389
PNEUMOTHORAX TRAUMATIC (Injury, poisoning and procedural complications) | 0/375 | 1/389
PRESYNCOPE (Nervous system disorders) | 1/375 | 0/389
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0/375 | 2/389
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0/375 | 1/389
PYREXIA (Respiratory, thoracic and mediastinal disorders) | 1/375 | 0/389
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/375 | 1/389
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1/375 | 0/389
RENAL FAILURE (Renal and urinary disorders) | 0/375 | 1/389
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1/375 | 1/389
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1/375 | 0/389
SHOCK (Vascular disorders) | 1/375 | 0/389
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1/375 | 0/389
SYNCOPE (Nervous system disorders) | 1/375 | 0/389
TESTICULAR CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/375 | 1/389
THROMBOSIS (Vascular disorders) | 1/375 | 0/389
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0/375 | 1/389
URINARY TRACT INFECTION (Infections and infestations) | 0/375 | 1/389
URTICARIA (Skin and subcutaneous tissue disorders) | 1/375 | 0/0
UVEITIS (Eye disorders) | 1/375 | 0/0
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1/375 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole (N=375) | Placebo (N=389)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 13
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 6 | 10
ANAEMIA (Blood and lymphatic system disorders) | 0 | 6
CONSTIPATION (Gastrointestinal disorders) | 10 | 15
CYSTITIS (Infections and infestations) | 0 | 6
DIARRHOEA (Gastrointestinal disorders) | 7 | 0
DIZZINESS (Nervous system disorders) | 6 | 5
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 8
HEADACHE (Nervous system disorders) | 8 | 11
HYPERTENSION (Vascular disorders) | 6 | 7
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 7
INSOMNIA (Psychiatric disorders) | 0 | 9
NAUSEA (Gastrointestinal disorders) | 11 | 10
PHLEBITIS (Vascular disorders) | 9 | 0
PYREXIA (Skin and subcutaneous tissue disorders) | 17 | 14
URINARY TRACT INFECTION (Infections and infestations) | 7 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AstraZeneca shall have a period of 30 days from receipt of the proposed final manuscript for any publication or other disclosure to review it and may within such time require that submission for publication or disclosure of the manuscript be delayed.